CLINICAL TRIAL: NCT04383288
Title: Prospective Observational Study of the Expression of ABCB1 / P-glycoprotein as a Factor for the Biological Stratification of Non-metastatic Osteosarcoma of the Extremities
Brief Title: ABCB1/P-glycoprotein Expression Influence on Non-metastatic Osteosarcoma of the Extremities
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Other Study IDs: GEIS-33
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — DNA from peripheral blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Overexpression of ABCB1 / P-glycoprotein. Poor response: If there is overexpression of ABCB1 / P-glycoprotein and poor response to induction treatment, in many sites ifosfamide at high doses and MTP-PE (Muramyl tripeptide phosphatidylethanolamine), is incorporated in addition to adriamycin.
  BEFORE SURGERY TREATMENT:
  Methotrexate: 12g/m2 (3 cycles) Cisplatinum: 120mg/m2 (3 cycles) Doxorubicin: ADM (Adriamycin) 75mg/m2 (3 cycles)
  AFTER SURGERY TREATMENT for poor responder patients with positive P-GLYCOPROTEIN Methotrexate 12g/m2; Cisplatinum 120mg/m2; Doxorubicin 90mg/m2 ifosfamide 15g/m2 MEPACT 2 mg/m2 twice a week for the first 3 months the weekly for the next 6 months (total length treatment 44 weeks)
  All the product are used as commercial formulation
  Other Names:
  Methotrexate Cisplatinum doxorubicin ifosfamide mifamurtide
- Overexpression of ABCB1 / P-glycoprotein. Good response: If there is overexpression of ABCB1 / P-glycoprotein and a good response to induction treatment, in many centers the option of additional administration of methotrexate, CDDP (Cisplatinum) and adriamycin will be chosen.
  BEFORE SURGERY TREATMENT:
  Methotrexate: 12g/m2 (3 cycles) Cisplatinum: 120mg/m2 (3 cycles) Doxorubicin: ADM 75mg/m2 (3 cycles)
  AFTER SURGERY TREATMENT for good responder patients with positive P-GLYCOPROTEIN Methotrexate 12g/m2 (10 Cycles) Cisplatinum 120mg/m2; Doxorubicin 90mg/m2 MEPACT 2 mg/m2 twice a week for the first 3 months the weekly for the next 6 months (total length treatment 44 weeks)
  All the product are used as commercial formulation
  Other Names:
  Methotrexate Cisplatinum doxorubicin ifosfamide mifamurtide
- No overexpression of ABCB1 / P-glycoprotein: If there is no overexpression of ABCB1 / P-glycoprotein, the administration of methotrexate, adriamycin and cisplatin will be chosen in many sites.
  BEFORE SURGERY TREATMENT:
  Methotrexate: 12g/m2 (3 cycles) Cisplatinum: 120mg/m2 (3 cycles) Doxorubicin: ADM 75mg/m2 (3 cycles)
  AFTER SURGERY TREATMENT:
  Methotrexate 12g/m2 (10 cycles) Cisplatinum 120mg/m2; Doxorubicin 90mg/m2
  Total length 34 weeks
  All the product are used as commercial formulation
  Other Names:
  methotrexate cisplatin doxorubicine

SUMMARY:
Post-authorization, observational, multicenter and prospective study in patients between 2 and 30 years old diagnosed with non-metastatic high-grade osteosarcoma of the extremities.

All patients included in the study will receive the initial neoadjuvant treatment prescribed by the doctor of each center, according to standard practice (involving methotrexate, cisplatin, and adriamycin). This initial treatment precedes surgical treatment.

After surgical treatment, the histological response to neoadjuvant chemotherapy will be evaluated. The histological response to primary chemotherapy will be expressed as a percentage of tumor necrosis. In the case of tumor necrosis above 90% the patient is defined as a "good responder" in case of a lower percentage as a "poor responder".

As an adjuvant treatment, the following options may be given according to standard practice in each center:

1. - If there is overexpression of ABCB1 / P-glycoprotein and poor response to induction treatment, in many sites ifosfamide at high doses and MTP-PE, is incorporated in addition to adriamycin.
2. - If there is overexpression of ABCB1 / P-glycoprotein and a good response to induction treatment, in many centers the option of additional administration of methotrexate, CDDP and adriamycin will be chosen.
3. - If there is no overexpression of ABCB1 / P-glycoprotein, the administration of methotrexate, adriamycin and cisplatin will be chosen in many sites.

In some sites they will consider the non-administration of MTP-PE or the non-administration of high doses of ifosfamide. And, in some hospitals, they will consider administering MTP-PE to all patients.

DETAILED DESCRIPTION:
The Primary objective is:

- Disease-free survival measured as a 5-year rate in patients with localized osteosarcoma treated, according to standard practice, with all the drugs currently registered for the treatment of non-metastatic osteosarcoma (methotrexate, cisplatin, adriamycin, ifosfamide, MTP-PE), according to ABCB1 / P-glycoprotein expression.

The Secondary objectives are:

* Evaluate overall survival in a homogeneous population of patients with non-metastatic osteosarcoma.
* Disease-free survival at 2 and 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed histological diagnosis of high-grade osteosarcoma of the extremities.
2. Age: from 2 to 30 years old.
3. Localized disease (metastasis skip accepted).
4. Normal liver, kidney and spinal function.
5. Ventricular ejection fraction of 50%.
6. Absence of previous surgical treatments or chemotherapy for osteosarcoma.
7. Interval between histological diagnosis and initiation of chemotherapy not exceeding 4 weeks.
8. Signing of the consent form to participate in the study.

Exclusion Criteria:

1. Presence of lung metastases on chest CT or in other locations.
2. Parosteal, periosteal, or secondary osteosarcoma.
3. Contraindications of the medications prescribed in the protocol.
4. Pregnant or lactating.
5. Mental or social conditions that do not guarantee adequate adherence to the protocol.
6. Not having an adequate understanding of study participation.

Ages: 12 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients from 2 to 30 years old diagnosed with non-metastatic high-grade osteosarcoma of the extremities.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Overall Survival | The patients will be followed in term of Overall Survival, for all the study period (expected average: 7 years)
  The Overall Survival will be evaluated at the end of the study period (5 enrollment years and 2 years - minimum- follow-up from the last enrolled patient)

SECONDARY OUTCOMES:
Events free survival | After 2 and 3 years from the start of study
  The events free survival will be evaluated by means of interim analysis after 2 and 3 years from the start of study. A further evaluation will be performed at the end of enrollment and after 2 years form the last enrolled patient.

CONTACTS AND LOCATIONS:
Overall Officials: Óscar Gallego, Dr., Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Luis Gros, Dr., Principal Investigator — Hospital Vall d'Hebron
Locations (17):
- Spain (17):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infantil Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Palmerini E, Meazza C, Tamburini A, Marquez-Vega C, Bisogno G, Fagioli F, Ferraresi V, Milano GM, Coccoli L, Rubio-San-Simon A, Gallego O, Llinares Riestra ME, Manzitti C, Mora J, Vaz-Salgado MA, Luksch R, Mata C, Pierini M, Carretta E, Cesari M, Paioli A, Marrari A, Scotlandi K, Serra M, Asaftei SD, Gambarotti M, Picci P, Ferrari S, Valverde C, Ibrahim T, Broto JM. Is There a Role for Mifamurtide in Nonmetastatic High-Grade Osteosarcoma? Results From the Italian Sarcoma Group (ISG/OS-2) and Spanish Sarcoma Group (GEIS-33) Trials. J Clin Oncol. 2025 Oct;43(28):3113-3122. doi: 10.1200/JCO-25-00210. Epub 2025 Aug 18. PMID 40825172